CLINICAL TRIAL: NCT02545959
Title: Intrathecal Rituximab in Progressive Multiple Sclerosis
Acronym: EFFRITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Dr Mickaël BONNAN, MD, Centre Hospitalier de PAU
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHPAU2014/01
Record Dates: First submitted 2015-09-07; First posted 2015-09-10 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis, Chronic Progressive; Nervous System Diseases
Keywords: Intrathecal Rituximab; intrathecal chemotherapy; cerebrospinal fluid; lumbar puncture; Physiological Effects of Drugs; Rituximab
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Nervous System Diseases | interventions — Rituximab; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): receive a single pulse of methylprednisolone IV (120mg)
  Interventions: Drug: methylprednisolone IV
- Rituximab IT group (Experimental): receive a single intrathecal infusion of rituximab (with IV methylprednisolone 120mg to avoid side effect)
  Interventions: Drug: Rituximab IT; Drug: methylprednisolone IV
- Rituximab IT + IV group (Experimental): receive Rituximab IT as previous and Rituximab IV (375mg/m2) the same day
  Interventions: Drug: Rituximab IT; Drug: methylprednisolone IV; Drug: Rituximab IV

INTERVENTIONS:
Drug: Rituximab IT — CSF injection of intrathecal rituximab (20mg)
  Other Names: intrathecal rituximab (Mabthera)
  Arms: Rituximab IT + IV group; Rituximab IT group
Drug: methylprednisolone IV — blood infusion of methylprednisolone IV (120mg)
  Other Names: Solumedrol
Drug: Rituximab IV — Blood infusion of rituximab (375mg/m2)
  Other Names: Mabthera
  Arms: Rituximab IT + IV group

SUMMARY:
The goal of investigators is to study the kinetics of action of a single dose of intrathecally-infused rituximab upon cerebro-spinal fluid (CSF) biological targets in progressive MS patients. Various markers of central nervous system inflammation (osteopontin, Tumor Necrosis Factor α, IgG secretion) and neurodegeneration (neurofilament) are studied at multiple time-points, assuming that a definitive action upon CSF biological targets would be strongly predictive of a delayed clinical action.

DETAILED DESCRIPTION:
• Background : Multiple sclerosis (MS) is the most frequent inflammatory disorder leading to impairment in young people. Although many drugs are now available to treat the early relapsing-remitting phase of MS (RR-MS), impairment is mostly linked to the secondary progressive phase of MS. Since no treatment proved to efficiently prevent or cure this progressive phase, treating this phase remains challenging. In fact, progressive phase is associated with a fence-ringed intrathecal compartmentalization of inflammation, leading to the unavailability of most immunosuppressive drugs. As a consequence, investigators here propose to shift the therapeutic paradigm in MS to a new paradigm based on intrathecal infusion of monoclonal antibodies (mAb) aimed at eradicate intrathecal inflammation. Rituximab is a mAb targeting CD20+ B-lymphocytes. Positive results in RR-MS were obtained after blood infusion of rituximab, but results were negative in progressive MS, probably due to the very low penetration of the blood brain barrier. Since intrathecal rituximab is already used in central nervous system (CNS) lymphomas, investigators propose to use it this way in progressive MS.

• Detailed description : An optimal dosage of rituximab for intrathecal infusion was choose using data already obtained in CNS lymphoma, acknowledging that 20mg offers the higher dosage with good tolerance profile. In order to isolate rituximab effect, a control group is treated by steroids since steroids are required before rituximab infusion. Moreover, B-lymphocytes depletion in CSF will probably be transient, as it is when rituximab is infused in blood. Assuming that CSF B-cells repopulation may be facilitated by peripheral B-cells, a group was assigned to receive also blood infusion of rituximab. CSF will be examined at multiple time points to assess the time frame of biological effect obtained in CSF.

Three groups of 4 patients are treated at day 0 :

1. Control group : receive a single pulse of intravenous (IV) methylprednisolone (120mg) ;
2. Rituximab intrathecal (IT) group : receive a single intrathecal infusion of rituximab (with IV methylprednisolone 120mg to avoid side effect) ;
3. Rituximab IT + IV group : receive same as previous and IV rituximab (375mg/m2) the same day.

CSF and blood will be drawn for study at day 0 (before treatment), day 4, day 21 and day 180. B- lymphocytes monitoring in blood will be also be done at day 365. A detailed clinical monitoring (walking time, nine hole peg test, Expanded Disability Status Score (EDSS), Symbol Digit Modalities Test (SDMT), fatigue intensity scale) will be done at each time point from day 0 to 365, assessing tolerance and clinical effect. MRI will be done at screening, months 6 and 12.

* Primary outcome : Change from baseline in Osteopontin level in CSF at day 4. CSF level is expected to normalize.
* Secondary outcomes: Biological outcomes in CSF (IgG synthesis, Tumor Necrosis Factor α, neurofilament) at day 4; delay to regain pre-therapeutic levels of biological targets in CSF (day 21, day 180) ; clinical data (walking time, nine hole peg test, Expanded Disability Status Score (EDSS), Symbol Digit Modalities Test (SDMT), fatigue intensity scale) at each time point, and brain MRI volumetry at day 180 and day 365.
* Study design : monocentric prospective randomized open clinical trial (phase II).
* Eligibility criteria:

Inclusion criteria:

* Age ≥45 years,
* male or female ;
* Secondary or primary progressive MS, in progressive phase since >2 years ;
* EDSS ≥6.0 ;
* Absence of alternative therapy.

Exclusion criteria:

* Relapsing-remitting phase of MS;
* Contraindication to MRI, lumbar puncture, Trendelenburg position ;
* Active infection or immunosuppressive state or treatment (actual or less than 6 months);
* Earlier treatment with rituximab;
* Dementia or severe psychiatric disorder.

  * Arm number or label and arm type :

experimental = Rituximab IT and Rituximab IT + IV groups ; comparator = Control group (methylprednisolone).

* Interventions : Three groups of 4 patients are treated at day 0 : 1) Control group : receive a single pulse of IV methylprednisolone (120mg) ; 2) Rituximab IT group : receive a single intrathecal infusion of rituximab (with IV methylprednisolone 120mg to avoid side effect) ; 3) Rituximab IT + IV group : receive same as previous and IV rituximab (375mg/m2) the same day.
* Number of subjects : 4 per group, with a total of 12 patients.
* Statistical analysis : target sample size was estimated based on an expected outcome of complete clearance of intrathecal inflammation from CNS compartment, which expected to normalize biological markers of CSF inflammation. The estimated size was 6.8 in treatment group and 3.4 in control group. We decided to include respectively 8 and 4 patients in treatment and control groups. Analyses will be performed at the 0.05 global level of significance, risk alpha = 0.05 and risk beta = 0.10. We will use the SAS 9.1.3 software.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years, male or female ;
* Secondary or primary progressive MS, in progressive phase since >2 years ;
* EDSS ≥6.0 ;
* Absence of alternative therapy.

Exclusion Criteria:

* Relapsing-remitting phase of MS;
* Contraindication to MRI, lumbar puncture, Trendelenburg position ;
* Active infection or immunosuppressive state or treatment (actual or less than 6 months);
* Earlier treatment with rituximab;
* Dementia or severe psychiatric disorder.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Change in osteopontin level in CSF | at day 4, day 21, day 180

SECONDARY OUTCOMES:
Change in Tumor Necrosis Factor alpha level in CSF | day 4, day 21, day 180
Change in IgG synthesis in CSF | day 4, day 21, day 180
Change in neurofilament level in CSF | day 4, day 21, day 180

OTHER OUTCOMES:
Change in clinical parameters | day 4, day 21, day 180, day 365
  Subjective appreciation and multiple clinical scales (walking time, nine hole peg test, EDSS, SDMT, Fatigue Intensity Scale)
Brain volume atrophy | day 180, day 365
  Percent change in total brain volume (SIENA)

CONTACTS AND LOCATIONS:
Overall Officials: Mickael Bonnan, MD, Principal Investigator — CH Pau
Locations (1):
- Centre hospitalier F. Mitterrand (CH Pau), Pau, France

REFERENCES:
- [Background] Bonnan M, Ferrari S, Bertandeau E, Demasles S, Krim E, Miquel M, Barroso B. Intrathecal rituximab therapy in multiple sclerosis: review of evidence supporting the need for future trials. Curr Drug Targets. 2014;15(13):1205-14. doi: 10.2174/1389450115666141029234644. PMID 25355180
- [Background] Bonnan M. Intrathecal immune reset in multiple sclerosis: exploring a new concept. Med Hypotheses. 2014 Mar;82(3):300-9. doi: 10.1016/j.mehy.2013.12.015. Epub 2013 Dec 31. PMID 24417802